CLINICAL TRIAL: NCT01624896
Title: The China PEACE (Patient-centered Evaluative Assessment of Cardiac Events) Prospective Study of Coronary Catheterization and Percutaneous Coronary Intervention
Brief Title: China PEACE-Retrospective CathPCI Study
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Sponsor
Other Study IDs: WSGY-201202025-2
Record Dates: First submitted 2012-06-17; First posted 2012-06-21 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Coronary heart disease (CHD) is one of the leading causes of mortality and morbidity. PCI, as a well-proved and booming measure in CHD management, is invasive and of high cost, however the knowledge about the real-life PCI use in China is limited. Within a nation-wide and regional representative probability sample of hospitals in China, 14,000 CAG/PCI inpatient cases will be sampled randomly from 2001 to 2011. The sampled medical records will be reviewed and abstracted in the national coordinating centre, in order to evaluate the treatment pattern, outcomes, and cost for PCI, during the past decade. Basic data and innovative evidence will accelerate evidence-based clinical practice and policy making, and improve patients outcomes in future finally.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a major concern in public health globally, as well as in China, and remarkable variations of resources available and health system performance have been noted. Relatively limited information is available about how evidence-based therapies are incorporated appropriately into routine clinical practice. In addition, little information is available about the magnitude and quality of PCI, which has developed rapidly during the past several decades. Practical and applied knowledge from large unselected population is needed to guide practice and policy for quality improvement and cost reduction.

To investigate the treatment pattern and outcomes of PCI during the past decade in China, using a stratified two-stage cluster sampling design, from 70 sampled hospitals, 7,000 CAG/PCI cases will be selected in 2011, and 3,500 in 2001 and 2006 separately. Photocopies of the 14,000 medical records of CAG/PCI cases will be sent to the national coordinating centre. Demographic characteristics, medical history, clinical features, diagnostic tests, medications, procedures, and in-hospital outcomes of patients will be abstracted by well trained professional abstractors. By characterizing differences in patients' features, comparing the use of medications and procedures, and examining the in-hospital outcomes, we'll define the gaps between clinical practice and guidelines, as well as the disparities across different regions and hospitals, to evaluated the treatment pattern and outcomes in the last decade in China. New knowledge will be generated about PCI management all over China, to provide evidence for policy-making and clinical guidelines, and to improve patients prognosis in future finally.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients undergoing a diagnostic cardiac catheterization and/or percutaneous coronary intervention (PCI) for coronary lesions.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Using a stratified two-stage cluster sampling design, 70 hospitals will be selected from different regions in China, and 7,000 PCI inpatient cases will be selected in 2011, and 3,500 in 2001 and 2006 separately, from these sample hospitals.
Sampling Method: Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Severe complications after PCI | Duration of hospital stay, an expected average of 1 week
  Composite of severe complications after PCI including coronary artery dissection, coronary spasm, acute coronary artery occlusion, thrombosis, acute myocardial infarction, emergent coronary artery bypass graft, death

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, M.D., Ph.D., Principal Investigator — China National Center for Cardiovascular Diseases; Harlan M Krumholz, M.D., S.M., Principal Investigator — Yale University

REFERENCES:
- [Derived] Li J, Dharmarajan K, Li X, Lin Z, Normand SL, Krumholz HM, Jiang L; China PEACE Collaborative Group. Protocol for the China PEACE (Patient-centered Evaluative Assessment of Cardiac Events) retrospective study of coronary catheterisation and percutaneous coronary intervention. BMJ Open. 2014 Mar 7;4(3):e004595. doi: 10.1136/bmjopen-2013-004595. PMID 24607563